CLINICAL TRIAL: NCT00784290
Title: Phase I/II Study of TSU-68 for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taiho132070
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — orantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Orantinib
  Interventions: Drug: Orantinib (TSU-68)

INTERVENTIONS:
Drug: Orantinib (TSU-68) — 200 or 400 mg bid day 1～day 28 cycle until progression or unacceptable toxicity develops

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Orantinib, an oral tyrosine kinase inhibitor of vascular endothelial growth factor receptor-2, platelet-derived growth factor receptor, and fibroblast growth factor receptor, in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
As HCC is a highly vascular tumor, a number of antiangiogenic agents have been tested for the treatment of HCC. Orantinib is an orally administered, small-molecule, multiple receptor tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor-2 (VEGFR-2), platelet-derived growth factor receptor (PDGFR), and fibroblast growth factor receptor (FGFR). Phase I studies that have been conducted in Japan for patients with solid tumors recommended a dosage of 400 mg bid. As a potent antiangiogenic agent, Orantinib is also expected to be effective against HCC. However, because most HCC patients have accompanying liver cirrhosis or hepatitis, its safety must be reevaluated in the presence of liver function impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-74
* PS 0-2
* Patients who did not respond to surgery, RFA, TAE, chemotherapy, or radiotherapy
* Chid-Pugh A or B
* At least one measurable lesion by RECIST criteria

Exclusion Criteria:

* Large amount of pleural effusion or ascites
* Esophageal varices
* Simultaneously active double cancer

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-09; Primary Completion 2010-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Step 1(Phase I) Safety | During chemotherapy
Step 2(Phase II) Response rate(RR) | Until progression

SECONDARY OUTCOMES:
Step 1(Phase I) Response rate(RR) | Until progression
Step 2(Phase II) Safety | During chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Masao Omata, M.D., Study Chair — Yamanashi Prefectural Central Hospital
Locations (1):
- Chiba University Hospital, Inohana Chuo-ku Chiba, Chiba, Japan

REFERENCES:
- [Derived] Enooku K, Tateishi R, Kanai F, Kondo Y, Masuzaki R, Goto T, Shiina S, Yoshida H, Omata M, Koike K. Evaluation of molecular targeted cancer drug by changes in tumor marker doubling times. J Gastroenterol. 2012 Jan;47(1):71-8. doi: 10.1007/s00535-011-0462-2. Epub 2011 Sep 21. PMID 21935635
- [Derived] Kanai F, Yoshida H, Tateishi R, Sato S, Kawabe T, Obi S, Kondo Y, Taniguchi M, Tagawa K, Ikeda M, Morizane C, Okusaka T, Arioka H, Shiina S, Omata M. A phase I/II trial of the oral antiangiogenic agent TSU-68 in patients with advanced hepatocellular carcinoma. Cancer Chemother Pharmacol. 2011 Feb;67(2):315-24. doi: 10.1007/s00280-010-1320-2. PMID 20390419